CLINICAL TRIAL: NCT01452542
Title: A Pilot, Phase 1, Single-site, Single-dose, Randomized, Open-label, Two-treatment, Two-sequence, Four-period Replicated Crossover Study Evaluating the Within-subject Pharmacokinetic Variability and Relative Bioavailability of the Phase 3 and Common Blend Formulations of Eliglustat in Healthy Adult Subjects.
Brief Title: A Phase I Study of the Pharmacokinetic Variability and Relative Bioavailability of the Phase 3 and Common Blend Formulations of Eliglustat in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GZGD03811
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteer
Keywords: Genz-112638
MeSH Terms: interventions — eliglustat; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Participants will receive a single oral dose of the following two study treatments under fasting conditions, in accordance with a randomly allocated treatment sequence: three 50-mg Phase 3 capsules of eliglustat (Reference Treatment [R]) or one 150-mg common blend capsule of eliglustat (Test Treatment [T]) according to the following treatment sequence: TRTR, with a 7-day washout between dosing in each period.
  Interventions: Drug: Eliglustat, common blend proposed commercial formulation; Drug: Eliglustat, Phase 3 capsule formulation
- Sequence 2 (Experimental): Participants will receive a single oral dose of the following two study treatments under fasting conditions, in accordance with a randomly allocated treatment sequence: three 50-mg Phase 3 capsules of eliglustat (Reference Treatment [R]) or one 150-mg common blend capsule of eliglustat (Test Treatment [T]) according to the following treatment sequence: RTRT, with a 7-day washout between dosing in each period.
  Interventions: Drug: Eliglustat, common blend proposed commercial formulation; Drug: Eliglustat, Phase 3 capsule formulation

INTERVENTIONS:
Drug: Eliglustat, common blend proposed commercial formulation — All participants will receive a single oral 150-mg dose of the common blend proposed commercial formulation of eliglustat, administered as one 150-mg strength capsule (Treatment T), on 2 separate dosing occasions.
  Other Names: Genz-112638
Drug: Eliglustat, Phase 3 capsule formulation — All participants will receive a single oral 150-mg dose of the Phase 3 capsule formulation of eliglustat, administered as three 50-mg strength capsules (Treatment R), on 2 separate dosing occasions.
  Other Names: Genz-112638

SUMMARY:
The primary objective of this pilot study is to determine the within-subject pharmacokinetic (PK) variability and relative bioavailability of single oral 150-mg doses of eliglustat administered as the Phase 3 formulation (3x50-mg capsules) and the common blend proposed commercial formulation (1x150-mg capsule) in healthy adult subjects, which will be used to plan and support the design of a subsequent bioequivalence study.

DETAILED DESCRIPTION:
This will be a single-site, single-dose, randomized, open-label, two-treatment, two-sequence, four-period replicated crossover study in healthy adult subjects. The study will comprise a screening period, four treatment periods with a 7-day washout between dosing in each period, and a safety follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* The subject is willing and able to provide signed informed consent.
* The subject is a male or female in good general health and between 18 and 45 years of age, inclusive.
* The subject has a body weight of 50 to 100 kg (110 to 220 lb) with a body mass index (BMI) ≤32 kg/m2 at screening.
* The subject's physical examination, laboratory, vital sign, and ECG test results are within normal limits at screening and Day -3 or, if abnormal, are not considered clinically significant in the opinion of the Investigator.
* The subject has been a non-smoker for at least 6 months prior to the time of providing informed consent, and is willing and able to abstain from smoking (and use of other forms of nicotine) until completion of the safety follow-up visit.
* The subject has not used drugs of abuse for at least 6 months prior to Day -1 and is willing and able to abstain from using drugs of abuse until completion of the safety follow-up visit.
* The subject is willing and able to abstain from alcohol for 48 hours prior to the first dose of study drug until completion of the safety follow-up visit.
* The subject is willing and able to abstain from grapefruit or star fruit products for 72 hours prior to the first dose of study drug until completion of the safety follow-up visit.
* The subject, if a female of childbearing potential, has a documented negative pregnancy test at screening and Day 1, and is willing to use a medically accepted form of contraception (as defined in the protocol) from screening until 30 days after the last dose of study drug. A woman of childbearing potential is defined as any female who has not been amenorrheic for at least 2 years or has not undergone a hysterectomy or surgical sterilization.

Exclusion Criteria:

* The subject is classified as a CYP2D6 poor metabolizer (or an indeterminate metabolizer with neither allele known to be active) or CYP2D6 ultra-rapid metabolizer (or an indeterminate metabolizer where one allele is known to correspond to ultra-rapid metabolism) based on results of CYP2D6 genotyping performed at screening. (Note: Prior CYP2D6 genotyping results may be used for the purpose of determining study eligibility if a copy of the laboratory report is available and the genotyping results can be interpreted with the same classification system used by the study reference laboratory.)
* The subject has a digestive disorder, including malabsorption, gastroenteritis, pancreatitis, gastroesophageal reflux disease, or inflammatory bowel disease (including Crohn's disease), or any other digestive disorder which, in the opinion of the Investigator, may affect oral bioavailability (e.g., clinically significant constipation, diverticulitis, or irritable bowel syndrome).
* The subject has had a GI surgical procedure that might affect drug transit time, (e.g., cholecystectomy, GI bypass surgery, partial or total gastrectomy, or small bowel resection).
* The subject has any of the following: Clinically significant coronary artery disease including history of myocardial infarction or ongoing signs or symptoms consistent with cardiac ischemia or heart failure; clinically significant arrhythmias or conduction defect such as 2nd or 3rd degree AV block, complete bundle branch block, prolonged QTc interval (e.g., repeated demonstration of a QTc interval ≥450 msec), or sustained ventricular tachycardia.
* The subject has any other clinically significant organic disease, including cardiovascular, renal, hepatic, GI, pulmonary, neurologic, endocrine, metabolic, or psychiatric disease, or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, precludes participation in the trial.
* The subject has received treatment with an inducer of CYP3A4 within 30 days prior to the first dose of study drug.
* The subject has received treatment with an inhibitor of CYP3A4 or CYP2D6 within 30 days prior to the first dose of study drug.
* The subject has received an immunization within 30 days prior to the first dose of study drug.
* The subject has received an investigational product within 60 days prior to the first dose of study drug or plans to receive any other investigational product at any time during the course of this study.
* The subject has received any other prescription or non-prescription medication (with the exception of nonprescription-strength ibuprofen and acetaminophen, topical non-steroidal preparations, and topical hydrocortisone (up to 1% strength)) or dietary or herbal supplement within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug, without the approval of both the Investigator and Sponsor.
* The subject has a history of drug allergies that are clinically significant in the opinion of the Investigator (e.g., significant rash or hives).
* The subject has a screening laboratory test result above the upper limit of normal for any of the following liver function tests: aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyltransferase (GGT), and total bilirubin.
* The subject tests positive for human immunodeficiency virus (HIV) antibody, hepatitis C antibody, or hepatitis B surface antigen at screening.
* The subject tests positive for urine drugs of abuse, urine alcohol, or urine cotinine at screening.
* The subject donated blood or blood products within 30 days prior to providing informed consent.
* The subject's schedule or travel plans prevent the completion of all required visits.
* The subject is scheduled for inpatient hospitalization, including elective surgery (inpatient or outpatient), during the study.
* The subject has a history of cancer, with the exception of basal cell carcinoma.
* The subject, if female, is pregnant or lactating.
* The subject, in the opinion of the Investigator, is unable to adhere to the requirements of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Eliglustat plasma concentration over time | Plasma concentration-time data will be obtained pre-dose (within 30 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, 48, and 72 hours after dosing in each treatment period.

SECONDARY OUTCOMES:
Area under the plasma concentration time curve (AUC) from time zero to the last time with a quantifiable concentration (AUClast) of eliglustat | Pre-dose (within 30 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, 48, and 72 hours after dosing in each treatment period.
Area under the concentration time curve (AUC) from time zero extrapolated to infinity (AUC0-∞) of eliglustat | Pre-dose (within 30 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, 48, and 72 hours after dosing in each treatment period.
Maximum observed eliglustat plasma concentration (Cmax) | Pre-dose (within 30 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, 48, and 72 hours after dosing in each treatment period.
Time to maximum observed plasma concentration (Tmax) | Pre-dose (within 30 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, 48, and 72 hours after dosing in each treatment period.
Apparent volume of distribution (Vz/F) of eliglustat | Pre-dose (within 30 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, 48, and 72 hours after dosing in each treatment period.
Apparent clearance (CL/F) of eliglustat | Pre-dose (within 30 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, 48, and 72 hours after dosing in each treatment period.
Terminal elimination rate constant (λz) of eliglustat | Pre-dose (within 30 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, 48, and 72 hours after dosing in each treatment period.
Terminal elimination half-life (t1/2) of eliglustat | Pre-dose (within 30 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 18, 24, 36, 48, and 72 hours after dosing in each treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- PPD Phase 1 Unit, Austin, Texas, United States